CLINICAL TRIAL: NCT04274816
Title: Releasing the Brakes on CD8+ T Cells in the Melanoma Sentinel Lymph Node by Pre-operative Local Administration of Low-dose Anti-CTLA-4 (Tremelimumab)
Brief Title: Intradermal Injection of Anti-CTLA-4 in Patients With Stage I/II Melanoma
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: A.J.M. van den Eertwegh (Other)
Responsible Party: Sponsor-Investigator, A.J.M. van den Eertwegh, Principal Investigator, Amsterdam UMC, location VUmc
Organization: Amsterdam UMC, location VUmc (Other)
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: 2011-000139-10
Record Dates: First submitted 2020-02-06; First posted 2020-02-18 (Actual); Last update posted 2020-02-18 (Actual); Status verified 2020-02

CONDITIONS: Cutaneous Melanoma
Keywords: Stage I-II melanoma; Anti-CTLA-4; Immunotherapy; Neoadjuvant
MeSH Terms: conditions — Melanoma | interventions — tremelimumab; Ipilimumab

STUDY DESIGN:
Intervention Model Description: Seven days before undergoing a SNB, clinical stage I/II melanoma patients will be treated with an intradermal injection of tremelimumab, around the excision site of the primary tumor. Escalating doses of 2, 5, 10, or 20 mg of tremelimumab will be given (3 patients per dose level with an expansion at the optimal dose level with an additional 5 patients).
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- Tremelimumab (Experimental): Intradermal injection of tremelimumab at the primary melanoma excision site, 7 days prior to sentinel node biopsy (SNB), with escalating doses of 2, 5, 10 or 20 mg tremelimumab (3 patients per dose level with an expansion at the optimal dose level with an additional 5 patients).
  Interventions: Drug: Tremelimumab

INTERVENTIONS:
Drug: Tremelimumab — Intradermal injection of tremelimumab 7 days prior to sentinel node biopsy, with escalating doses of 2, 5, 10 or 20 mg tremelimumab (3 patients per dose level with an expansion at the optimal dose level with an additional 5 patients).
  Other Names: Anti-CTLA-4

SUMMARY:
This study evaluates the clinical safety and tolerability, and the immunological effects of local intradermal injection of tremelimumab in patients with clinical stage I/II melanoma patients undergoing a sentinel node biopsy (SNB). Patients will be treated by local intradermal injections around the excision site of the primary tumor with escalating doses of 2, 5, 10 or 20 mg tremelimumab.

DETAILED DESCRIPTION:
Although of limited therapeutic value, the SLN procedure has proven a useful prognostic tool for the assessment of melanoma relapse and mortality risk. Moreover, the SLN is of great value for the assessment of immunological interventions for melanoma. Since early melanoma development is accompanied by impaired immune effector functions primarily in the SLN, there is a strong rationale for therapeutic immune modulation of the SLN aimed at strengthening cellular immune functions.

The investigator now propose a phase I dose escalation study to administer intradermally a single clinical dose of tremelimumab/anti-CTLA-4 locally at the primary tumor excision site of patients with clinical stage I/II melanoma. Such a single local administration aimed at conditioning of the SLN should allow for the use of relatively low anti-CTLA-4 dosages without excess risk of autoimmune effects.

ELIGIBILITY:
Inclusion Criteria:

* Age ≥ 18 years
* Clinical stage I/II melanoma patients, planned to undergo a sentinel lymph node biopsy (SNB)
* ECOG performance status 0 or 1
* White blood count (WBC) ≥ 3 x10^9/L
* Platelet count ≥ 100 x10^9/L
* Hemoglobin ≥ 6.5 mmol/L
* Serum creatinine ≤ 2.5 x ULN
* Total serum bilirubin, AST, ALT and LDH ≤ 2x ULN

Exclusion Criteria:

* Non-oncology vaccine therapy used for prevention of infectious diseases (up-to) 4 weeks prior and/r 8 weeks after any dose of tremelimumab
* Prior treatment with a CD137 agonist or CTLA-4 inhibitor or agonist
* Uncontrolled infectious disease including negative testing for HIV, HBV, HCV
* Autoimmune disease

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 13 (Actual)
Dates: Start 2012-07-10 (Actual); Primary Completion 2014-02-27 (Actual); Study Completion 2014-02-27 (Actual)

PRIMARY OUTCOMES:
Number of participants with adverse events as assessed by CTCAE V3.0 | From the time of injection until 28 days after injection of tremelimumab
  The descriptions and grading scales of CTCAE V 3.0 will be utilized for all toxicity reporting
Change in frequency of immune cell populations (compared to baseline) assessed by immune monitoring through flow cytometry, | 7 days after the intradermal injection of tremelimumab
  Blood samples and sentinel lymph node material will be collected and then analyzed by flow cytometry. Changes in frequency of tumor-specific T-cells, Tregs and dendritic subsets will be assesess and compared to baseline (time of the injection of the intradermal injection)
Change in activation status of immune cell populations (compared to baseline) assessed by immune monitoring through flow cytometry, | 7 days after the intradermal injection of tremelimumab
  Blood samples and sentinel lymph node material will be collected and then analyzed by flow cytometry. Changes in expression level of surface antigens for tumor-specific T-cells, Tregs and dendritic subsets are analyzed and compared to baseline (time of injection of tremelimumab)

CONTACTS AND LOCATIONS:
Overall Officials: Tanja D de Gruijl, Principal Investigator — Amsterdam UMC, location VUmc; Alfons JM van den Eertwegh, Principal Investigator — Amsterdam UMC, location VUmc

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Derived] van Pul KM, Notohardjo JCL, Fransen MF, Koster BD, Stam AGM, Chondronasiou D, Lougheed SM, Bakker J, Kandiah V, van den Tol MP, Jooss K, Vuylsteke RJCLM, van den Eertwegh AJM, de Gruijl TD. Local delivery of low-dose anti-CTLA-4 to the melanoma lymphatic basin leads to systemic Treg reduction and effector T cell activation. Sci Immunol. 2022 Jul 15;7(73):eabn8097. doi: 10.1126/sciimmunol.abn8097. Epub 2022 Jul 15. PMID 35857579